CLINICAL TRIAL: NCT07001553
Title: Understanding the Dietary Adjustments Following GLP-1 Agonist Treatment: The GLaD Feasibility Study
Brief Title: Understanding Acute Dietary Changes After GLP-1 Agonist Treatment: The GLaD Feasibility Study
Acronym: GLaD
Status: Recruiting | Type: Observational
Sponsor: Australian Catholic University (Other)
Collaborators: St Vincent's Hospital Melbourne (Other); The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-4090H
Record Dates: First submitted 2025-05-22; First posted 2025-06-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Type 2 Diabetes Mellitus (T2DM)
Keywords: dietary behaviours; psychosocial health
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Weight management: Prescribed GLP-1 agonist therapy primarily for weight management
- Type 2 diabetes: Prescribed GLP-1 agonist therapy primarily for glycemic management

SUMMARY:
An observational study of those who have been prescribed a GLP-1 agonist therapy (yet to commence), for either weight or diabetes management, and are willing to complete dietary records and questionnaires of behaviour and psychosocial health.

DETAILED DESCRIPTION:
Forty individuals (20 for weight management, 20 for diabetes management) living in Australia who have been prescribed a GLP-1 agonist (no previous prescription or no use in the previous 6 months) will be recruited to participate over the initial 3 months of their treatment. Assessments will occur remotely (online) at baseline, 2 weeks, 1 month and 3 months. Optional body composition assessments will be provided at baseline and 3 months for those based in Melbourne, Australia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+ years old
* Intending to commence a prescription for a GLP-1 agonist (may be dual agonist, i.e. Ozempic, Trulicity, Monjaro, or Saxenda) medication, with no use in the previous 6 months
* The primary reason for commencing the medication will be for diabetes or weight management
* Willing to participate in dietary recall and questionnaires

Exclusion Criteria:

* Aged under 18 years,
* used a GLP-1 agonist medication in the previous 6 months,
* unwilling or unable to provide dietary recalls
* non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals living in Australia who are intending to commence a GLP-1 prescription
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | 4 months
  The rate of recruitment and the retention rate of participants completing the dietary assessment measures.

SECONDARY OUTCOMES:
Energy intake | baseline, 2 weeks, 1 month, 3 months
  Assessed using Intake24 records for at least 2 days per timepoint
Medication symptomology | baseline, 1 month, 3 months
  Incidence of self-reported side effects
Medication use | baseline, 1 month, 3 months
  Dosage

OTHER OUTCOMES:
Patient perspectives | 3 months
  Qualitative interview after end of the observation period
Macronutrient intake | baseline, 2 weeks, 1 month, 3 months
  Proportion of carbohdyrate, fat, protein, alcohol and fibre intake assessed through dietary records
Diet quality | baseline, 2 weeks, 1 month, 3 months
  Assessed using Healthy Eating Index for Australian adults (HEIFA) from diet records (Intake24)
Meal timing | baseline, 2 weeks, 1 month, 3 months
  Daily eating window and meal timing
Medication use | baseline, 1 month, 3 months
  Timing of medication use
Retrospective subjective appetite | baseline, 1 month, 3 months
  Assessed using adaptive visual analogue scales with appetite questions as per Flint et al 2020 and used by Ravussin et al 2025, scored between 0 to 100, with a higher score meaning higher appetite ratings
Treatment self-regulation | baseline, 1 month, 3 months
  Assessed using Treatment Self-regulation Questionnaire, 15 questions which are scored between 1 (not at all) and 7 (completely true) in response to questions
Food cravings | baseline, 1 month, 3 months
  Assessed using Control of Eating Questionnaire (COEQ), a 21 questionnaire survey with a 0-100 scale where higher responses indicate higher severity of food cravings.
Internalisation of weight bias | baseline, 1 month, 3 months
  Assessed using Weight Bias Internalisation Scale-Modified (WBIS-M), which includes 11 questions that are answered on a 1 (strongly disagree) to 7 (strongly agree) scale, noting that 2 questions are reverse scored.
Intuitive eating | baseline, 1 month, 3 months
  Assessed using Intuitive Eating Scale 3 (IES-3), including 12 questions with options from 1 (strongly disagree) to 5 (strongly agree) where the higher total score indicates higher intuitive eating (Tykla et al, Appetite, 2024)
Health-related quality of life | baseline, 1 month, 3 months
  Assessed using Short Form-36 (SF-36) questionnaire, where 36 questions are asked regarding the previous 4 weeks. Questions are given a score between 0 to 100 depending, and the overall score is the average of all questions.
Well being | baseline, 1 month, 3 months
  Quality of life assessed using WHO-5 well being index, including 5 questions scored from 0 (none of the time) to 5 (all of the time), where a higher total score indicates better quality of life.
Binge eating | baseline, 1 month, 3 months
  Assessed using Binge eating scale, which includes 16 questions. The total score ranges from 0 to 46, with higher scores correlating with more frequent and severe binge eating behaviours.
Disordered eating behaviours | baseline, 1 month, 3 months
  Assessed using Eating Disorders Examination Questionnaire (EDEQ) 6.0, using 28 questions which are scored on 4 sub-scales and a global score is generated as an average of the 4 sub-scales. A higher score indicates greater disordered eating behaviours.
Physical activity | baseline, 1 month, 3 months
  Assessed using International Physical Activity Questionnaire (long), which is 27 questions which asks duration (minutes) and frequency (days) of physical activity measured in domains of: 1) Job-related; 2) Transportation; 3) Housework, house maintenance, caring for family; 4) Recreation, sport, and leisure-time; and 5) Time spent sitting. An overall score is calculated using responses to all questions, where a higher score equates to greater physical activity.
Dietary changes | baseline, 3 months
  Assessed using Australian Eating Survey Food Frequency Questionnaire (FFQ), which has 120-item with 15 supplementary questions. The FFQ is designed to collect information about dietary intake over the participants previous 3 months.
Micronutrient intake | baseline, 2 weeks, 1 month, 3 months
  Proportion of micronutrient intake (i.e. including but not limited to sodium, calcium, iron, zinc, vitamins, etc) assessed through dietary records

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn B Parr, PhD, Principal Investigator — Australian Catholic University
Locations (1):
- Australian Catholic University, Fitzroy, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the corresponding author for a period of 36 months from publication, upon reasonable request for academic use. The data will not be made publically available, as it contains information that could compromise research participant consent.
Supporting Information: Study Protocol, SAP
Time Frame: 36 months from date of publication
Access Criteria: Reasonable requests of data for academic use will be considered. Requests can be made to the corresponding author of the publication. Data will not be made publicly available as it contains information that could compromise research participant consent.